CLINICAL TRIAL: NCT02799654
Title: Non-Interventional Post Market Clinical Follow-up Study Excia T® Cementless EBRA Study
Brief Title: Excia T Cementless EBRA Study
Status: Withdrawn | Type: Observational
Why Stopped: Change of organizational circumstances.
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1612
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Arthritis, Degenerative; Arthritis, Rheumatoid; Hip Fractures; Femur Head Necrosis
Keywords: Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Hip Fractures; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this Post Market Clinical Follow-up Study (PMCF Study), the short-term clinical and radiological results of the cementless Excia T® prosthesis in routine clinical use shall be assessed and the migration taking place in the first 24 months evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Written patient consent to study participation
* Age > 18 years
* Indication for primary THA with cementless Excia T® stem

Exclusion Criteria:

* Pregnancy
* THA after fracture
* Rheumatoid arthritis
* Systemic disorders, treated with Cortisone or other pharmaceuticals, potentially compromising the bone quality
* Patient physically or mentally not able to follow the postoperative examination routine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for cementless primary Total Hip Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Subsidence over time of Excia T® stem (EBRA-FCA) | discharge (approx. 1 week postop), 3, 12 and 24 months postoperative
  The subsidence of the Excia T stem will be measured with Ein-Bild-Röntgen-Analysis Femoral Component Analysis (EBRA-FCA). EBRA allows a non-invasive measurement of routinely taken A/P radiographs. Necessary is a series of at least four x-rays that can be read by the EBRA software.
  The whole implant must be visible on the A/P x-ray, as well as the greater and lesser trochanter.
  Subsidence shall be measured on the follow-up x-rays in comparison to the discharge x-rays.

SECONDARY OUTCOMES:
Clinical Results over time (Harris Hip Score) | preoperative, discharge (approx. 1 week postop), 3, 12 and 24 months postoperative
  The clinical assessment will be done with the Harris Hip Score (HHS)
Quality of Life over time (EQ-5D-5L) | preoperative, discharge (approx. 1 week postop), 3, 12 and 24 months postoperative
  The generic patient reported outcome score EQ-5D-5L will be used for the assessment of quality of life.
Osteolysis over time (localized bone resorption) | 3, 12 and 24 months postoperative
  radiological evaluation will be done according to the (A/P) Gruen zones
Radiolucent lines over time | 3, 12 and 24 months postoperative
  radiological evaluation will be done according to the (A/P) Gruen zones: ≤1mm, 1-2mm, ≥2mm
Cortical thinning | 3, 12 and 24 months postoperative
  radiological evaluation will be done according to the (A/P) Gruen zones
Hypertrophy | 3, 12 and 24 months postoperative
  radiological evaluation will be done according to the (A/P) Gruen zones
Mechanical Alignment over time | discharge (approx. 1 week postop), 3, 12 and 24 months postoperative
  any change of the A/P implant angle (varus / valgus alignment) as assessed with EBRA-FCA will be evaluated
Adverse Events / Serious Adverse Events | until 24 months postoperative
  Rates of Adverse Events / Serious Adverse Events are recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. med. E. Mayr, Celle, Germany

IPD SHARING:
Plan to Share IPD: No